CLINICAL TRIAL: NCT02600871
Title: Skin and Soft Tissue Infection (SSTI) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20150722H
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-02

CONDITIONS: Skin Diseases, Infectious; Soft Tissue Infections
Keywords: Abscess; Antiseptic; Provodine; Povidone-Iodine
MeSH Terms: conditions — Skin Diseases, Infectious; Soft Tissue Infections; Abscess | interventions — Povidone-Iodine; Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provodine (Experimental): Provodine patients will have standard care including incision and drainage. The contents of 1 packet of Provodine applied with a Q-tip to the walls and floor of the abscess cavity. The contents of a 2nd packet will be applied to the surrounding skin within 5 cm around the incision.
  Provodine patients will return within 48-72 hours for a follow-up visit, have the packing removed and the contents of the packet reapplied to the abscess cavity and surrounding skin.
  Provodine patients will be instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They will wash their hands with soap and water, pat dry, and apply the contents of 1 packet of Provodine to dorsum and palmar aspects of hands and fingers and rub together for 1 minute. They will apply the contents of a 2nd packet to the abscess cavity, and a 3rd packet to the surrounding skin. They will be then rinse their hands with water, pat dry, and cover the wound with 4x4 gauze.
  Interventions: Drug: Provodine; Procedure: Incision and Drainage
- Standard Care (Active Comparator): Standard care patients will have standard care including incision and drainage.
  Standard care patients will return within 48-72 hours for a follow-up visit and have the packing removed.
  Standard care patients will be instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They will cover wound with 4x4 gauze and wash hands with soap and water for 1 minute.
  Interventions: Procedure: Incision and Drainage

INTERVENTIONS:
Drug: Provodine
  Other Names: Povidone-Iodine
  Arms: Provodine
Procedure: Incision and Drainage

SUMMARY:
The purpose of this study is to determine if the use Provodine as an antiseptic and hand wash once daily for at least 7 days will have better healing, better health outcomes, fewer treatment failures and fewer infections themselves and among their household contacts than those who do not use Provodine.

DETAILED DESCRIPTION:
Patients who meet criteria for the study will be enrolled by a convenience sample and randomized to a treatment group. Each patient will have a demographic data sheet completed by one of the study investigators or research associates. The data sheet will include contact information, age, gender, ethnicity, location of the abscess, measured length and width of palpable fluctuance and induration, measured length and width of surrounding cellulitis, presence or absence of fever, and previous medical history (including history of prior skin abscesses.) Assignment to a treatment group will be by blocked randomization.

All enrolled patients will be provided with an informed consent document and an overview of the study. Baseline measurements including size of abscess (measured by ruler of palpable fluctuance and induration) and maximal diameter of the largest area of cellulitis will be recorded. Providers will outline the area of palpable fluctuance with an Aspen skin marker and delineate the surrounding area of cellulitis with a dotted line to establish baseline surface area of wound. All patients will have standard care including incision and drainage and wound culture of the abscess cavity. All patients will receive local anesthesia and additional pain management will be left to the discretion of the treating provider. Providers will make a linear incision over the length of palpable fluctuance and induration. The provider will explore the wound cavity and break apart any loculations to allow for adequate drainage of purulent discharge. The provider will obtain wound cultures and irrigate with normal saline until clear irrigation fluid drains from cavity. Swabs will be sub-cultured on blood agar plates and grown overnight for bacterial identification and antibiotic susceptibility testing.

Patients randomized to Provodine will have the abscess cavity and surrounding skin gently painted with Provodine solution. The contents of one foil packet of Provodine will be applied with a Q-tip to the walls and floor of the abscess cavity. The contents of a second foil packet will be applied to the surrounding skin within 5 cm around the incision.

The abscess cavity of both groups will be gently packed with ¼ inch plain gauze strips and the wound will be covered with 4x4 gauze and secured with tape. Patients will be instructed to leave the wound packing in place and change the outer dressing once a day until they return at 48-72 hours for their first wound recheck.

Several studies have shown that there is no clinical benefit to antibiotics in the routine management of uncomplicated abscesses. Patients with uncomplicated abscesses (defined as palpable abscess < 5 cm in a healthy patient with no history of diabetes, HIV, IVDA or immunocompromised state who has no systemic signs of infection) will not be treated with antibiotics. Patients who do not meet these criteria will be treated with antibiotics at the discretion of the provider.

A study investigator will evaluate the patient in the emergency department or clinic within 48- 72 hours for the initial follow up visit and the packing will be removed. Patients randomized to Provodine will have the contents of the foil packet reapplied to the walls of the abscess cavity and surrounding skin. Data that will be collected on initial recheck include presence or absence of fever, purulent drainage, erythema, and pain, as well as presence of new skin lesions. A new lesion is defined as a new abscess, pustule, carbuncle, or furuncle at least 5 cm away from the initial wound. Lesions within 5 cm of initial wound will be considered failures of the initial abscess treatment.

Study investigators will also record compliance with intervention and side effects. Compliance will be assessed by measuring the amount of opened foil packets and by patient report. The cure rate, as measured by the absence of fever, pain, erythema and purulent discharge, will be recorded as well as the overall assessment by the provider if wound is improving, unchanged, or clinically worsened.

Wound management will be left up to the discretion of the treating provider, but further incision and drainage, wound repacking and antibiotic use will be reserved for patients determined to be not clinically improving or getting worse and will be considered a treatment failure. Outcomes including clinical cure, rate of new lesion development in patients and HCs, and therapeutic changes to clinical management will be recorded.

After the packing is removed, all patients will be instructed to cleanse the abscess at home by soaking in water once a day and gently patting the wound dry. Patients will follow specific instructions for wound management once a day after washing.

After cleansing and drying the abscess, the patients randomized to the Provodine arm will wash their hands with soap and water, pat dry, and apply the contents of one foil packet of Provodine to dorsum and palmar aspects of hands and fingers and rub hands and fingers together for one minute to ensure all skin distal to the wrist is covered. They will then apply the contents of a second foil packet to the walls and floor of the abscess cavity using a Q tip applicator. The patient will then apply a third foil packet of Provodine to the skin surrounding the abscess within 5 cm diameter of the wound using a separate Q tip. After applying Provodine to the abscess and surrounding skin, they will be then gently rinse their hands with water, pat hands dry, and cover the wound with a 4x4 gauze dressing.

The patient will also be instructed to keep a sealable bag of empty Provodine foil packets to assess compliance at follow up visits.

Patients randomized to standard care will cover wound with 4x4 gauze dressing and wash hands with soap and water for one minute. Patients will be instructed to continue to perform once daily cleansing/treatments until they are seen for their second wound recheck or until wound cavity has closed.

The patient will return for a 2nd visit between 7 and 10 days for a second wound recheck. Data that will be collected will be the same as on initial recheck including the presence or absence of fever, purulent drainage, erythema, and pain, as well as presence of new skin abscesses in the patient or HCs.

Study investigators will also record compliance with intervention and side effects. Compliance will be assessed by measuring the amount of opened foil packets and by patient report. The cure rate, as measured by the absence of fever, pain, erythema and purulent discharge, will be recorded. Wound management will again be left up to the discretion of the treating provider, but further incision and drainage, wound repacking and antibiotic use will be encouraged only for patients determined to be not clinically improving or getting worse and will again be considered a treatment failure. Outcomes including clinical cure, reinfection, rate of new lesion development, and therapeutic changes to clinical management will be recorded.

Patients will be called at home at 30 days to assess for treatment failures requiring additional intervention and new lesion development in patients and their HCs.

Outcomes include rate of clinical cure rate of initial abscess and rate of new lesion development. Therapeutic changes (e.g., addition of new antibiotics or additional incision and drainage), or unplanned health care encounters for the skin infection (e.g., urgent care visits, emergent care visits, or hospital admissions) will be considered treatment failures. Fisher's exact test will be used to compare outcomes between groups.

Continuously distributed outcomes will be summarized with the sample size, mean, standard deviation, median, minimum and maximum, and categorical outcomes will be summarized with frequencies and percentages. The number screened, the number of screen failures by reason, and the number randomized, and the number lost to follow-up by reason and the number completing the study by treatment group will be tabulated. Treatment groups will be contrasted with regard to cure (yes, no), new lesions (yes, no), and infections (yes, no) with Fisher's Exact tests. Adverse events, if any, will be listed by treatment group and case number and indicators of seriousness (serious, not serious), severity (mild, moderate, severe), and relation to the treatment (related to the treatment, unknown but not related to the treatment). All statistical testing will be two-sided with a significance level of 5%. The sample size was not derived from a statistical power calculation but was motivated by the pilot nature of this study. SAS Version 9.4 for Windows or R will be used throughout.

ELIGIBILITY:
Inclusion Criteria:

* Skin abscess
* Treatment requiring incision and drainage

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Homeless, incarcerated, or living in a group home
* Abscess on the face or breast
* Abscess requiring surgical drainage in the operating room or requiring admission to the hospital
* Intravenous drug users
* Previous enrollment in this study
* Documented history of iodine sensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, San Antonio, Texas, United States

REFERENCES:
- [Background] Labreche MJ, Lee GC, Attridge RT, Mortensen EM, Koeller J, Du LC, Nyren NR, Trevino LB, Trevino SB, Pena J, Mann MW, Munoz A, Marcos Y, Rocha G, Koretsky S, Esparza S, Finnie M, Dallas SD, Parchman ML, Frei CR. Treatment failure and costs in patients with methicillin-resistant Staphylococcus aureus (MRSA) skin and soft tissue infections: a South Texas Ambulatory Research Network (STARNet) study. J Am Board Fam Med. 2013 Sep-Oct;26(5):508-17. doi: 10.3122/jabfm.2013.05.120247. PMID 24004702
- [Background] Schmitz GR, Bruner D, Pitotti R, Olderog C, Livengood T, Williams J, Huebner K, Lightfoot J, Ritz B, Bates C, Schmitz M, Mete M, Deye G. Randomized controlled trial of trimethoprim-sulfamethoxazole for uncomplicated skin abscesses in patients at risk for community-associated methicillin-resistant Staphylococcus aureus infection. Ann Emerg Med. 2010 Sep;56(3):283-7. doi: 10.1016/j.annemergmed.2010.03.002. Epub 2010 Mar 26. PMID 20346539
- [Background] Duong M, Markwell S, Peter J, Barenkamp S. Randomized, controlled trial of antibiotics in the management of community-acquired skin abscesses in the pediatric patient. Ann Emerg Med. 2010 May;55(5):401-7. doi: 10.1016/j.annemergmed.2009.03.014. Epub 2009 May 5. PMID 19409657

RESULTS

PARTICIPANT FLOW:
Groups:
- Provodine: Provodine patients had standard care including incision and drainage. The contents of 1 packet of Provodine were applied with a Q-tip to the walls and floor of the abscess cavity. The contents of a 2nd packet were applied to the surrounding skin within 5 cm around the incision.
  Provodine patients returned at 48-72 hours for a follow-up visit, had the packing removed and the contents of the packet reapplied to the abscess cavity and surrounding skin.
  Provodine patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They washed their hands with soap and water, patted dry, and applied the contents of 1 packet of Provodine to dorsum and palmar aspects of hands and fingers and rubbed together for 1 minute. They applied the contents of a 2nd packet to the abscess cavity, and a 3rd packet to the surrounding skin. They rinsed their hands with water, patted dry, and cover ed the wound with 4x4 gauze.
- Standard Care: Standard care patients had standard care including incision and drainage.
  Standard care patients returned at 48-72 hours for a follow-up visit and had the packing removed.
  Standard care patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They covered wound with 4x4 gauze and washed hands with soap and water for 1 minute.
Period: Overall Study
Arm/Group | Provodine | Standard Care
Started | 52 | 49
Completed | 39 (51 subjects completed the 7-10 day follow up 39 subjects completed the 30-day follow up) | 39 (45 subjects completed the 7-10 day follow up 39 subjects completed the 30-day follow up)
Not Completed | 13 | 10
Not completed — Lost to Follow-up | 13 | 10

BASELINE CHARACTERISTICS:
Groups:
- Provodine: Provodine patients had standard care including incision and drainage. The contents of 1 packet of Provodine applied with a Q-tip to the walls and floor of the abscess cavity. Contents of a 2nd packet were applied to the surrounding skin within 5 cm around the incision.
  Provodine patients returned at 48-72 hours for a follow-up visit, had the packing removed and the contents of the packet reapplied to the abscess cavity and surrounding skin.
  Provodine patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They washed their hands with soap and water, patted dry, and applied the contents of 1 packet of Provodine to dorsum and palmar aspects of hands and fingers and rubbed together for 1 minute. They applied the contents of a 2nd packet to the abscess cavity, and a 3rd packet to the surrounding skin. They rinsed their hands with water, patted dry, and covered the wound with 4x4 gauze.
- Standard Care: Standard care patients had standard care including incision and drainage.
  Standard care patients returned at 48-72 hours for a follow-up visit and have the packing removed.
  Standard care patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They covered the wound with 4x4 gauze and washed hands with soap and water for 1 minute.
- Total: Total of all reporting groups
Arm/Group | Provodine | Standard Care | Total
Number analyzed (Participants) | 52 | 49 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.33 (14.82) | 41.76 (13.57) | 41.53 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 33 | 30 | 63
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 9 | 10 | 19
  White | 5 | 9 | 14
  Black or African American | 9 | 3 | 12
  Other | 29 | 27 | 56
Abscess location [Count of Participants; unit: Participants]
  Trunk | 15 | 12 | 27
  Extremity | 17 | 14 | 31
  Groin/Buttock | 14 | 10 | 24
  Axilla | 5 | 6 | 11
  Head and Neck | 6 | 5 | 11
Cellulitis [Median (Inter-Quartile Range); unit: cm^2] | 5 [1.25 to 12.5] | 5 [0 to 9] | 5 [0 to 10.13]
Abscess size [Median (Inter-Quartile Range); unit: cm^2] | 18 [8 to 27] | 12 [5 to 33] | 15 [7.3 to 28.5]
Culture results [Count of Participants; unit: Participants]
  MRSA | 17 | 17 | 34
  MSSA | 6 | 10 | 16
  Coag neg Staph | 7 | 11 | 18
  Streptococcus | 5 | 6 | 11
  No growth | 4 | 2 | 6
  Other | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Clinical Cure
Description: Clinical cure was defined as improvement in the initial wound with respect to a decrease in measured size, erythema, and purulent discharge. Wound management at the follow up visits was left up to the discretion of the treating provider, but additional interventions for patients not clinically improving or worsening were considered a lack of clinical cure.
Time Frame: 7-10 Days
Measure: Count of Participants; unit: Participants
Groups:
- Provodine: Provodine patients had standard care including incision and drainage. The contents of 1 packet of Provodine was applied with a Q-tip to the walls and floor of the abscess cavity. The contents of a 2nd packet were applied to the surrounding skin within 5 cm around the incision.
  Provodine patients returned at 48-72 hours for a follow-up visit, had the packing removed and the contents of the packet reapplied to the abscess cavity and surrounding skin.
  Provodine patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They washed their hands with soap and water, patted dry, and applied the contents of 1 packet of Provodine to dorsum and palmar aspects of hands and fingers and rubbed together for 1 minute. They applied the contents of a 2nd packet to the abscess cavity, and a 3rd packet to the surrounding skin. They rinsed their hands with water, patted dry, and covered the wound with 4x4 gauze.
- Standard Care: Standard care patients had standard care including incision and drainage.
  Standard care patients returned within 48-72 hours for a follow-up visit and had the packing removed.
  Standard care patients were instructed to cleanse the abscess at home by soaking in water once a day and patting the wound dry. They then covered wound with 4x4 gauze and washed hands with soap and water for 1 minute.
Arm/Group | Provodine | Standard Care
Number analyzed (Participants) | 51 | 46
Participants | 45 | 42
Statistical Analysis 1: Comparison: Provodine vs Standard Care; Test type: Superiority — The significance of variation in proportions with treatment (Provodine®, Control) was assessed with Fisher's Exact tests and variation in the mean with treatment was assessed with T-tests; p = 0.71, Fisher Exact

2. Secondary Outcome: Infection Rates of Household Contacts
Description: New lesions (abscess, pustule, carbuncle, or furuncle) that developed in household contacts of subjects within 30 days of enrollment
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Provodine | Standard Care
Number analyzed (Participants) | 39 | 39
Participants | 2 | 4

3. Secondary Outcome: Rate of New Lesion Development
Description: New lesions, defined as a new abscess, pustule, carbuncle, or furuncle at least 5cm away from the initial wound, that developed in the subject within 30 days of enrollment
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Provodine | Standard Care
Number analyzed (Participants) | 39 | 41
Participants | 8 | 8

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Provodine | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/49
Other Adverse Events (participants affected / at risk) | 31/52 | 13/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Provodine (N=52) | Standard Care (N=49)
Burning/pain (Skin and subcutaneous tissue disorders) | 18 (18) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (2)
Tape irritation (Skin and subcutaneous tissue disorders) | 7 (7) | 7 (7)
Skin irritation around wound (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chills (Infections and infestations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Decreased appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The low sample size of subjects was insufficient to perform a power calculation. Not all patients were compliant with hand washing and Provodine use. The 30-day follow phone call was self-reported, and not all subjects could be contacted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT02600871/Prot_SAP_000.pdf